CLINICAL TRIAL: NCT06691919
Title: Surgical vs Endoscopic Resection Of Walled Off Pancreatic Necrosis Using The Powered Endoscopic Debridement (PED) System - The SERPENT Trial
Brief Title: Surgical vs Endoscopic Resection of Walled Off Pancreatic Necrosis Using the Powered Endoscopic Debridement System
Acronym: SERPENT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Indiana University Health (Other)
Responsible Party: Principal Investigator, Abel Joseph, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 78066
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Necrosis; Pancreatitis
Keywords: Direct Endoscopy Necrosectomy; Transgastric Surgical Necrosectomy; Powered Endoscopic Debridement; Pancreatic Necrosis; Walled of Pancreatic Necrosis; Necrotizing Pancreatitis
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Pancreatitis

STUDY DESIGN:
Intervention Model Description: "Endoscopy" arm will receive direct endoscopic necrosectomy and "Surgery" arm will undergo transgastric surgical necrosectomy.
Masking Description: Biostatistician will be blinded to the study groups while performing final study analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Direct Endoscopic Necrosectomy (Experimental): Subjects randomized to the endoscopy arm will undergo direct endoscopic necrosectomy using the Powered Endoscopic Debridement System which has CE-Mark 613797 and FDA De Novo clearance in the United States (DEN200016).
  Interventions: Device: Direct Endoscopic Necrosectomy with Powered Endoscopic Debridement
- Transgastric Surgical Necrosectomy (Experimental): Patients randomized to the surgical arm will undergo open or minimally invasive (laparoscopic) transgastric surgical necrosectomy (SN). In either approach, the peritoneal cavity is entered to identify the stomach through which an anterior gastrotomy is made. The retrogastric necrosum is identified either using a finder needle or ultrasound and accessed through a posterior cystgastrostomy. Transgastric SN is then manually performed, and any cyst fluid fully evacuated. The anterior gastrotomy is then closed allowing any residual necrosis or pancreatic enzyme to efflux into the stomach and enter the upper GI tract. As with endoscopy, patients with retrogastric collections are observed for a sufficient period to ensure full maturation of the necrosum.
  Interventions: Procedure: Transgastric Surgical Necrosectomy

INTERVENTIONS:
Device: Direct Endoscopic Necrosectomy with Powered Endoscopic Debridement — Patients will first undergo endoscopic ultrasound-guided cystgastrostomy using an electrocautery-enhanced lumen apposing metallic stent to gain access to the necrosum. Direct Endoscopic Necrosectomy will be performed using the EndoRotor® NecroMax 6.0 PED Catheter which has an outer diameter of 5.1 mm and is compatible with endoscopes that have a working channel of ≥6.0 mm.
  Arms: Direct Endoscopic Necrosectomy
Procedure: Transgastric Surgical Necrosectomy — Patients randomized to the surgical arm will undergo open or minimally invasive (laparoscopic) transgastric SN with the aim of creating an ample size cystgastrostomy to perform a complete debridement. In either approach, the peritoneal cavity is entered to identify the stomach through which an anterior gastrotomy is made. The retrogastric necrosum is identified either using a finder needle or ultrasound and accessed through a posterior cystgastrostomy. Transgastric SN is then manually performed, and any cyst fluid fully evacuated. The anterior gastrotomy is then closed allowing any residual necrosis or pancreatic enzyme to efflux into the stomach and enter the upper GI tract. As with endoscopy, patients with retrogastric collections are observed for a sufficient period to ensure full maturation of the necrosum.
  Arms: Transgastric Surgical Necrosectomy

SUMMARY:
Goal:

The goal of this clinical trial is to compare the effectiveness and safety of two different but highly effective treatment approaches for walled-off necrosis (WON) resulting from severe acute pancreatitis.

Participant Population:

The study will involve adult patients experiencing symptomatic WON due to acute necrotizing pancreatitis.

Main Questions:

The main questions it aims to answer are:

1. Is "endoscopy" or direct endoscopic necrosectomy (DEN) with powered endoscopic debridement (PED) as effective as "surgery" or transgastric surgical necrosectomy (SN) in achieving clinical resolution of WON within six weeks after treatment?
2. What are the rates of complications, costs, hospital length of stay, procedure time, readmission, repeat procedures and overall patient satisfaction associated with DEN with PED compared to transgastric SN?

Comparison Group:

Researchers will compare the outcomes of patients receiving DEN with PED to those undergoing transgastric SN to see if there are significant differences in clinical success, rates of complications, and overall healthcare costs.

Participants Will:

1. Be randomly assigned to one of the two treatment groups (DEN with PED or transgastric SN).
2. Undergo the assigned treatment procedure based on their group.
3. Complete assessments before and after the procedure to evaluate clinical outcomes, hospital stay length, quality of life, and patient satisfaction.
4. Be monitored for adverse events or complications following the treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or greater.
* Patients with first episode of symptomatic WON+ due to acute pancreatitis (+Persistent fatigue, malaise, abdominal pain, gastric outlet obstruction, early satiety, fever, chills, jaundice, reduced appetite, persistent nausea/vomiting, steatorrhea)
* Patients who are candidates for surgical or endoscopic necrosectomy of WON as deemed by a multidisciplinary committee of HPB surgeons and therapeutic endoscopists.
* Patients who can tolerate repeat procedures.
* Subjects with the ability to understand the requirements of the study, who have provided written informed consent, and who are willing and able to return for the required follow-up assessments.

Exclusion Criteria:

* Documented untreated pseudoaneurysm within WON.
* Subject unable or unwilling to provide informed consent.
* Intervening gastric varices or unavoidable blood vessels within the WON access tract (visible using pre-procedural imaging).
* Coagulation disorders or anti-coagulant therapy which cannot be discontinued for the intervention to an absolute cardiac or vascular indication such as ACS, Stroke, Mechanical cardiovascular valves.
* Pregnant or lactating women or women of childbearing potential who do not employ a reliable method of contraception as judged by the Investigator, and/or are not willing to use reliable contraception for the duration of study participation.
* Patient is enrolled in another trial that could interfere with the endpoint analyses of this trial.
* Non-communicating pancreatic or extra-pancreatic fluid collections.
* Extensive abdominal surgical history due to peritoneal adhesions, prior open or recent operation during pancreatitis course, or remote gastric surgery that precludes a transgastric surgical cystgastrostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Treatment Success at 6 weeks after Debridement | From initial intervention to 6 weeks
  Clinical resolution is defined as clinical improvement of WON symptoms precluding the need for additional endoscopic or surgical interventions.
  AND Radiographic resolution defined as >70% reduction in WON on CT or MR imaging.

SECONDARY OUTCOMES:
Overall treatment success rate at end of 6-month follow-up from date of intervention | From initial intervention to the end of followup at 6 months
  Clinical resolution is defined as clinical improvement of WON symptoms precluding the need for additional endoscopic or surgical interventions after completion of 6-month follow-up.
  AND Radiographic resolution defined as >70% reduction in WON on CT or MR imaging after completion of 6-month follow-up.
Clinical improvement within 72 hours of debridement | From initial intervention to 72 hours after treatment
  Clinical improvement is defined according to the criteria used in the PANTER and TENSION trial. (8-10) "Clinical improvement" defined as: i. Improved function of at least two organ systems (i.e. circulatory, pulmonary, renal) according to the Investigator's medical judgement within 72 hours of the procedure, or; ii. At least 10% improvement of two out of three parameters of infection (i.e. C-reactive protein, leucocyte count or temperature) within 72 hours of the procedure.
  Deterioration of these parameters by other infectious causes (e.g.urinary tract infection) will be excluded.
Clinical Failure at 6 months | From initial intervention to the end of followup at 6 months
  Absence of clinical improvement or clinical deterioration
30-day mortality | From initial intervention to followup at 30 days
  Mortality occurring at 30 days after intervention
Overall total cost of care | From initial intervention to the end of followup at 6 months
  Cost of care per patient to achieve overall treatment success
Overall cost of care at 6 weeks | From initial intervention to followup at 6 weeks
  Cost of care per patient to achieve overall primary outcome
Percent reduction in WON collection volume (cm3) at 6-month follow-up | From initial intervention to the end of followup at 6 months
  Percent reduction in overall size of the WON collection volume (cm3) compared to pre-treatment CT or MR imaging.
Percent resolution of solid necrosum in patients with pre-and post-MR imaging at 6-month follow up | From initial intervention to the end of followup at 6 months
  Percent reduction in solid necrosis component of the WON collection volume (cm3) compared to pre-treatment MRI scan.
Post-procedural length of hospitalization (recovery time) | From index intervention to hospital discharge at 6 weeks
  Length of hospitalization from index intervention to hospital discharge
Readmissions | From initial intervention to the end of followup at 6 months
  Number of hospital readmissions due to disease or procedure-related symptoms or events.
Reintervention rates | From initial intervention to the end of followup at 6 months
  Need for endoscopic, radiological, or surgical intervention for additional drainage or necrotic debridement after the index intervention, excluding the follow-up procedure at 4-weeks for LAMS removal
Requirement of percutaneous drain | From initial intervention to the end of followup at 6 months
  Need for additional drainage with percutaneous drain
Total anesthesia duration | On day of intervention (1 day)
  Total duration of anesthesia of primary intervention
Procedure-related adverse events | From initial intervention to the end of followup at 6 months
  Any adverse event resulting from endoscopic intervention (yes/no)
Disease-related adverse events | From initial intervention to the end of followup at 6 months
  Any adverse event resulting from necrotizing pancreatitis
Patient satisfaction | From initial intervention to the end of followup at 6 months
  Patient satisfaction of primary intervention at 6 weeks post intervention graded on a visual analog scale (0-10)
Subject quality of life (QOL) | From initial intervention to the end of followup at 6 months
  Quality of life survey to participants at 6 month follow up. Patients will be asked to place a mark on a horizontal 10 cm line indicating his/her QoL from very poor to very good. The wording will be: "How would you rate your overall quality of life?". Higher score indicates very good quality of life and lower score indicates poor quality of life. The instrument is valid and has been used in clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Joo Ha Hwang, MD, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li AY, Bergquist JR, Visser BC. Necrosectomy in the Management of Necrotizing Pancreatitis. Adv Surg. 2021 Sep;55:231-250. doi: 10.1016/j.yasu.2021.05.016. No abstract available. PMID 34389094
- [Background] Onnekink AM, Boxhoorn L, Timmerhuis HC, Bac ST, Besselink MG, Boermeester MA, Bollen TL, Bosscha K, Bouwense SAW, Bruno MJ, van Brunschot S, Cappendijk VC, Consten ECJ, Dejong CH, Dijkgraaf MGW, van Eijck CHJ, Erkelens WG, van Goor H, van Grinsven J, Haveman JW, van Hooft JE, Jansen JM, van Lienden KP, Meijssen MAC, Nieuwenhuijs VB, Poley JW, Quispel R, de Ridder RJ, Romkens TEH, van Santvoort HC, Scheepers JJ, Schwartz MP, Seerden T, Spanier MBW, Straathof JWA, Timmer R, Venneman NG, Verdonk RC, Vleggaar FP, van Wanrooij RL, Witteman BJM, Fockens P, Voermans RP; Dutch Pancreatitis Study Group. Endoscopic Versus Surgical Step-Up Approach for Infected Necrotizing Pancreatitis (ExTENSION): Long-term Follow-up of a Randomized Trial. Gastroenterology. 2022 Sep;163(3):712-722.e14. doi: 10.1053/j.gastro.2022.05.015. Epub 2022 May 14. PMID 35580661
- [Background] Olsen GA, Schmidt PN, Novovic S, Hansen EF, Karstensen JG. Novel powered 5.0-mm endoscopic debridement catheter for endoscopic transmural necrosectomy of pancreatic walled-off necrosis: a case series of consecutive patients from a tertiary referral center (with video). Gastrointest Endosc. 2024 Feb;99(2):267-270. doi: 10.1016/j.gie.2023.10.044. Epub 2023 Oct 20. PMID 37865281
- [Background] Bang JY, Arnoletti JP, Holt BA, Sutton B, Hasan MK, Navaneethan U, Feranec N, Wilcox CM, Tharian B, Hawes RH, Varadarajulu S. An Endoscopic Transluminal Approach, Compared With Minimally Invasive Surgery, Reduces Complications and Costs for Patients With Necrotizing Pancreatitis. Gastroenterology. 2019 Mar;156(4):1027-1040.e3. doi: 10.1053/j.gastro.2018.11.031. Epub 2018 Nov 16. PMID 30452918
- [Background] van Brunschot S, van Grinsven J, van Santvoort HC, Bakker OJ, Besselink MG, Boermeester MA, Bollen TL, Bosscha K, Bouwense SA, Bruno MJ, Cappendijk VC, Consten EC, Dejong CH, van Eijck CH, Erkelens WG, van Goor H, van Grevenstein WMU, Haveman JW, Hofker SH, Jansen JM, Lameris JS, van Lienden KP, Meijssen MA, Mulder CJ, Nieuwenhuijs VB, Poley JW, Quispel R, de Ridder RJ, Romkens TE, Scheepers JJ, Schepers NJ, Schwartz MP, Seerden T, Spanier BWM, Straathof JWA, Strijker M, Timmer R, Venneman NG, Vleggaar FP, Voermans RP, Witteman BJ, Gooszen HG, Dijkgraaf MG, Fockens P; Dutch Pancreatitis Study Group. Endoscopic or surgical step-up approach for infected necrotising pancreatitis: a multicentre randomised trial. Lancet. 2018 Jan 6;391(10115):51-58. doi: 10.1016/S0140-6736(17)32404-2. Epub 2017 Nov 3. PMID 29108721
- [Background] Seifert H, Biermer M, Schmitt W, Jurgensen C, Will U, Gerlach R, Kreitmair C, Meining A, Wehrmann T, Rosch T. Transluminal endoscopic necrosectomy after acute pancreatitis: a multicentre study with long-term follow-up (the GEPARD Study). Gut. 2009 Sep;58(9):1260-6. doi: 10.1136/gut.2008.163733. Epub 2009 Mar 11. PMID 19282306
- [Background] Puli SR, Graumlich JF, Pamulaparthy SR, Kalva N. Endoscopic transmural necrosectomy for walled-off pancreatic necrosis: a systematic review and meta-analysis. Can J Gastroenterol Hepatol. 2014 Jan;28(1):50-3. doi: 10.1155/2014/539783. Epub 2013 Nov 8. PMID 24212912
- [Background] Worhunsky DJ, Qadan M, Dua MM, Park WG, Poultsides GA, Norton JA, Visser BC. Laparoscopic transgastric necrosectomy for the management of pancreatic necrosis. J Am Coll Surg. 2014 Oct;219(4):735-43. doi: 10.1016/j.jamcollsurg.2014.04.012. Epub 2014 May 29. PMID 25158913
- [Background] Fugazza A, Sethi A, Trindade AJ, Troncone E, Devlin J, Khashab MA, Vleggaar FP, Bogte A, Tarantino I, Deprez PH, Fabbri C, Aparicio JR, Fockens P, Voermans RP, Uwe W, Vanbiervliet G, Charachon A, Packey CD, Benias PC, El-Sherif Y, Paiji C, Ligresti D, Binda C, Martinez B, Correale L, Adler DG, Repici A, Anderloni A. International multicenter comprehensive analysis of adverse events associated with lumen-apposing metal stent placement for pancreatic fluid collection drainage. Gastrointest Endosc. 2020 Mar;91(3):574-583. doi: 10.1016/j.gie.2019.11.021. Epub 2019 Nov 20. PMID 31759037
- [Background] van der Wiel SE, Poley JW, Grubben MJAL, Bruno MJ, Koch AD. The EndoRotor, a novel tool for the endoscopic management of pancreatic necrosis. Endoscopy. 2018 Sep;50(9):E240-E241. doi: 10.1055/a-0628-6136. Epub 2018 Jun 19. No abstract available. PMID 29920619
- [Background] Maatman TK, McGuire SP, Flick KF, Madison MK, Al-Haddad MA, Bick BL, Ceppa EP, DeWitt JM, Easler JJ, Fogel EL, Gromski MA, House MG, Lehman GA, Nakeeb A, Schmidt CM, Sherman S, Watkins JL, Zyromski NJ. Outcomes in Endoscopic and Operative Transgastric Pancreatic Debridement. Ann Surg. 2021 Sep 1;274(3):516-523. doi: 10.1097/SLA.0000000000004997. PMID 34238810
- [Background] Stassen PMC, de Jonge PJF, Bruno MJ, Koch AD, Trindade AJ, Benias PC, Sejpal DV, Siddiqui UD, Chapman CG, Villa E, Tharian B, Inamdar S, Hwang JH, Barakat MT, Andalib I, Gaidhane M, Sarkar A, Shahid H, Tyberg A, Binmoeller K, Watson RR, Nett A, Schlag C, Abdelhafez M, Friedrich-Rust M, Schlachterman A, Chiang AL, Loren D, Kowalski T, Kahaleh M. Safety and efficacy of a novel resection system for direct endoscopic necrosectomy of walled-off pancreas necrosis: a prospective, international, multicenter trial. Gastrointest Endosc. 2022 Mar;95(3):471-479. doi: 10.1016/j.gie.2021.09.025. Epub 2021 Sep 22. PMID 34562471
- [Background] Bang JY, Lakhtakia S, Thakkar S, Buxbaum JL, Waxman I, Sutton B, Memon SF, Singh S, Basha J, Singh A, Navaneethan U, Hawes RH, Wilcox CM, Varadarajulu S; United States Pancreatic Disease Study Group. Upfront endoscopic necrosectomy or step-up endoscopic approach for infected necrotising pancreatitis (DESTIN): a single-blinded, multicentre, randomised trial. Lancet Gastroenterol Hepatol. 2024 Jan;9(1):22-33. doi: 10.1016/S2468-1253(23)00331-X. Epub 2023 Nov 18. PMID 37980922
- [Background] Driedger M, Zyromski NJ, Visser BC, Jester A, Sutherland FR, Nakeeb A, Dixon E, Dua MM, House MG, Worhunsky DJ, Munene G, Ball CG. Surgical Transgastric Necrosectomy for Necrotizing Pancreatitis: A Single-stage Procedure for Walled-off Pancreatic Necrosis. Ann Surg. 2020 Jan;271(1):163-168. doi: 10.1097/SLA.0000000000003048. PMID 30216220
- [Background] Bakker OJ, van Santvoort HC, van Brunschot S, Geskus RB, Besselink MG, Bollen TL, van Eijck CH, Fockens P, Hazebroek EJ, Nijmeijer RM, Poley JW, van Ramshorst B, Vleggaar FP, Boermeester MA, Gooszen HG, Weusten BL, Timmer R; Dutch Pancreatitis Study Group. Endoscopic transgastric vs surgical necrosectomy for infected necrotizing pancreatitis: a randomized trial. JAMA. 2012 Mar 14;307(10):1053-61. doi: 10.1001/jama.2012.276. PMID 22416101
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Tenner S, Baillie J, DeWitt J, Vege SS; American College of Gastroenterology. American College of Gastroenterology guideline: management of acute pancreatitis. Am J Gastroenterol. 2013 Sep;108(9):1400-15; 1416. doi: 10.1038/ajg.2013.218. Epub 2013 Jul 30. PMID 23896955
- [Background] Arvanitakis M, Dumonceau JM, Albert J, Badaoui A, Bali MA, Barthet M, Besselink M, Deviere J, Oliveira Ferreira A, Gyokeres T, Hritz I, Hucl T, Milashka M, Papanikolaou IS, Poley JW, Seewald S, Vanbiervliet G, van Lienden K, van Santvoort H, Voermans R, Delhaye M, van Hooft J. Endoscopic management of acute necrotizing pancreatitis: European Society of Gastrointestinal Endoscopy (ESGE) evidence-based multidisciplinary guidelines. Endoscopy. 2018 May;50(5):524-546. doi: 10.1055/a-0588-5365. Epub 2018 Apr 9. PMID 29631305
- [Background] Peery AF, Crockett SD, Barritt AS, Dellon ES, Eluri S, Gangarosa LM, Jensen ET, Lund JL, Pasricha S, Runge T, Schmidt M, Shaheen NJ, Sandler RS. Burden of Gastrointestinal, Liver, and Pancreatic Diseases in the United States. Gastroenterology. 2015 Dec;149(7):1731-1741.e3. doi: 10.1053/j.gastro.2015.08.045. Epub 2015 Aug 29. PMID 26327134
- [Background] Trikudanathan G, Wolbrink DRJ, van Santvoort HC, Mallery S, Freeman M, Besselink MG. Current Concepts in Severe Acute and Necrotizing Pancreatitis: An Evidence-Based Approach. Gastroenterology. 2019 May;156(7):1994-2007.e3. doi: 10.1053/j.gastro.2019.01.269. Epub 2019 Feb 15. PMID 30776347